CLINICAL TRIAL: NCT02220738
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ABT-957 in Subjects With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Brief Title: Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ABT-957 in Subjects With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow subject enrollment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-334
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — alicapistat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-957 (Experimental): ABT-957 administered twice-daily for 7 days
  Interventions: Drug: ABT-957
- Placebo (Placebo Comparator): Placebo administered twice-daily for 7 days
  Interventions: Other: Placebo for ABT-957

INTERVENTIONS:
Drug: ABT-957 — ABT-957 administered twice-daily for 7 days
  Arms: ABT-957
Other: Placebo for ABT-957 — Placebo for ABT-957 administered twice-daily for 7 days
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the safety, tolerability and pharmacokinetics of multiple doses of ABT-957 in subjects with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Meets the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria for probable Alzheimer's disease (AD);
* Has a Mini-Mental State Examination total score of 16 to 26;
* Has a Modified Hachinski Ischemia Scale score of ≤ 4;
* Is taking a stable dose of donepezil, galantamine or rivastigmine for at least 30 days;
* Has had a computerized tomography or magnetic resonance imaging. The scan must not show evidence for an alternative etiology for dementia;
* With the exception of a diagnosis of mild-to-moderate AD and the presence of stable medical conditions, is in general good health.

Exclusion Criteria:

* Positive screen for drugs of abuse, alcohol or cotinine;
* Females must not have positive results for pregnancy;
* Focal neurological signs on examination;
* Has a clinically significant abnormal value, in serum chemistry, hematology or urinalysis;
* History of any significant neurologic disease other than AD;
* History of head trauma, motor vehicle accident, concussion.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic evaluation of the two ABT-957 diastereomers | Day 7
  maximum observed plasma concentration (Cmax), time to Cmax (peak time, Tmax), plasma concentration at the end of the dosing interval (Ctrough), the area under the plasma concentration-time curve (AUC) during each dosing interval (AUC0-12 and AUC12-24)
Number of subjects with adverse events | Routinely for the duration of the study, about 7 months
  Subjects will be monitored for clinical and laboratory evidence of adverse events throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Nuno Mendonca, MD, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 129545, Glendale, California
  - Site Reference ID/Investigator# 129435, Orlando, Florida
  - Site Reference ID/Investigator# 129641, New York, New York
  - Site Reference ID/Investigator# 144825, Salt Lake City, Utah

REFERENCES:
- [Result] Lon HK, Mendonca N, Goss S, Othman AA, Locke C, Jin Z, Rendenbach-Mueller B. Pharmacokinetics, Safety, Tolerability, and Pharmacodynamics of Alicapistat, a Selective Inhibitor of Human Calpains 1 and 2 for the Treatment of Alzheimer Disease: An Overview of Phase 1 Studies. Clin Pharmacol Drug Dev. 2019 Apr;8(3):290-303. doi: 10.1002/cpdd.598. Epub 2018 Jul 27. PMID 30052328